CLINICAL TRIAL: NCT04247100
Title: A Pilot Study of a Randomized Sham-control Auricular TENS Unit Stimulation to Improve Symptoms Through Vagal Modulation in Pediatric Functional Gastrointestinal Disorders
Brief Title: A Study of Randomized Sham-control Auricular TENS Unit Stimulation in Pediatric Functional Gastrointestinal Disorders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ended prior to hitting the enrollment goal
Sponsor: Gisela Grotewold Chelimsky (Other)
Responsible Party: Sponsor-Investigator, Gisela Grotewold Chelimsky, Professor of Pediatrics, Virginia Commonwealth University
Organization: Virginia Commonwealth University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM20026558
Record Dates: First submitted 2020-01-22; First posted 2020-01-29 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Functional Gastrointestinal Disorders; Vagus Nerve Autonomic Disorder; Irritable Bowel Syndrome; Nausea; Dyspepsia
MeSH Terms: conditions — Gastrointestinal Diseases; Irritable Bowel Syndrome; Nausea; Dyspepsia | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: 30 participants will be enrolled in this double-blind sham control study. Fifteen participants will undergo sham stimulation for 4 weeks followed by active microstimulation for 4 weeks. The other 15 participants will have active microstimulation for all 8 weeks.
Who Masked: Participant, Care Provider
Masking Description: Participants will be sent home at baseline with a TENS unit and a sealed envelope with instructions for device settings. The envelope will contain instructions for either sham stimulation or active stimulation (unknown to the performing coordinator and participant). Both groups will receive a new device and another set of instructions from the study team at 4 weeks. It is possible and permitted that the performing study coordinator will become aware of which group the subject is in when checking in on the subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Stimulation (8) (Experimental): Participants will receive active auricular microstimulation via TENS unit for 8 weeks.
  Under guidance from the study team, participants will self-administer the TENS therapy for two 1-hour periods a day for 8 weeks.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- Sham Stimulation (4), Active (4) (Sham Comparator): Participants will receive sham therapy via inactive TENS unit for 4 weeks, followed by active auricular microstimulation via TENS for 4 weeks.
  Under guidance from the study team, participants will self-administer the TENS therapy for two 1-hour periods a day for 8 weeks (4 weeks of therapy with inactive TENS, 4 weeks with active TENS).
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS); Device: Sham Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — Active Transcutaneous Auricular Microstimulation delivered by TENS device
  Other Names: InTENSity Select Combo by Roscoe Medical
Device: Sham Transcutaneous Electrical Nerve Stimulation — Sham therapy will be delivered by applying the TENS device with non-conductive electrodes so that no microstimulation is delivered
  Other Names: InTENSity Select Combo by Roscoe Medical (Inactive)
  Arms: Sham Stimulation (4), Active (4)

SUMMARY:
The purpose of this study is to see if using a micro-current through a device called a TENS (Transcutaneous Electrical Nerve Stimulator) unit helps to improve functional gastrointestinal disorder (FGID) symptoms in children by stimulation of the vagus nerve. The study will compare two methods of stimulation to determine if there is a difference in the two methods.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 12-18 years old with chronic idiopathic nausea, function abdominal pain, dyspepsia and/or irritable bowel syndrome
* English Speaking

Exclusion Criteria:

* Patients who are unable to stand upright during the heart rate variability recording
* Patients with a known bleeding disorder
* Gastric or cardiac pacer or defibrillator
* Poor circulation in lower limbs
* Swollen or inflamed outer ear
* Epilepsy
* Abdominal or inguinal hernia
* Any unstable medical condition, such as renal disease, uncontrolled diabetes, etc.
* Requires new medication during the 8 weeks of the study that may affect gastrointestinal symptoms, vagal modulation or immune response
* Inability to answer questionnaires or report pain on a 0-10 visual analog scale.

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gisela Chelimsky, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kovacic K, Hainsworth K, Sood M, Chelimsky G, Unteutsch R, Nugent M, Simpson P, Miranda A. Neurostimulation for abdominal pain-related functional gastrointestinal disorders in adolescents: a randomised, double-blind, sham-controlled trial. Lancet Gastroenterol Hepatol. 2017 Oct;2(10):727-737. doi: 10.1016/S2468-1253(17)30253-4. Epub 2017 Aug 18. PMID 28826627
- [Background] Brock C, Brock B, Aziz Q, Moller HJ, Pfeiffer Jensen M, Drewes AM, Farmer AD. Transcutaneous cervical vagal nerve stimulation modulates cardiac vagal tone and tumor necrosis factor-alpha. Neurogastroenterol Motil. 2017 May;29(5). doi: 10.1111/nmo.12999. Epub 2016 Dec 12. PMID 27957782
- [Background] Ji RR, Xu ZZ, Gao YJ. Emerging targets in neuroinflammation-driven chronic pain. Nat Rev Drug Discov. 2014 Jul;13(7):533-48. doi: 10.1038/nrd4334. Epub 2014 Jun 20. PMID 24948120

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Stimulation (8): Participants will receive active auricular microstimulation via TENS unit for 8 weeks.
  Under guidance from the study team, participants will self-administer the TENS therapy for two 1-hour periods a day for 8 weeks.
  Transcutaneous Electrical Nerve Stimulation (TENS): Active Transcutaneous Auricular Microstimulation delivered by TENS device
- Sham Stimulation (4), Active (4): Participants will receive sham therapy via inactive TENS unit for 4 weeks, followed by active auricular microstimulation via TENS for 4 weeks.
  Under guidance from the study team, participants will self-administer the TENS therapy for two 1-hour periods a day for 8 weeks (4 weeks of therapy with inactive TENS, 4 weeks with active TENS).
  Transcutaneous Electrical Nerve Stimulation (TENS): Active Transcutaneous Auricular Microstimulation delivered by TENS device
  Sham Transcutaneous Electrical Nerve Stimulation: Sham therapy will be delivered by applying the TENS device with non-conductive electrodes so that no microstimulation is delivered
Period: Overall Study
Arm/Group | Active Stimulation (8) | Sham Stimulation (4), Active (4)
Started | 5 | 5
Completed | 4 | 4
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Stimulation (8) | Sham Stimulation (4), Active (4) | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Full Range); unit: years] | 16 [15 to 18] | 15.3 [13 to 16] | 15.8 [13 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Heart Rate Variability at 4 Weeks
Description: EKG tracing will be used to analyze Heart Rate Variability as an indirect measure of vagal nerve output and central autonomic control.
Time Frame: Assessed at baseline, week 4, and week 8. Change in baseline to week 4 is reported.
Measure: Mean (Standard Deviation); unit: milliseconds (ms)^2
Arm/Group | Active Stimulation (8) | Sham Stimulation (4), Active (4)
Number analyzed (Participants) | 4 | 4
milliseconds (ms)^2
  Standing | -639 (988) | -264 (244)
  Supine | 5360 (11500) | -5440 (9340)

2. Primary Outcome: Change in Heart Rate Variability at 8 Weeks
Description: as for outcome 1
Time Frame: Assessed at baseline, week 4, and week 8. Change in baseline to week 8 is reported.
Measure: Mean (Standard Deviation); unit: milliseconds (ms)^2
Arm/Group | Active Stimulation (8) | Sham Stimulation (4), Active (4)
Number analyzed (Participants) | 4 | 4
milliseconds (ms)^2
  Standing | -678 (1520) | -65.9 (613)
  Supine | 1640 (3750) | -8550 (11200)

3. Primary Outcome: Change in Mitochondrial Bioenergetics Measured by Basal Oxygen Consumption Rate at 4 Weeks (Basal Consumption)
Description: Blood draw will be tested for mitochondrial function by Seahorse assay, which measures Basal Oxygen Consumption Rate of live cells to provide insight into mitochondrial activity.
Time Frame: Assessed at baseline, week 4, and week 8. Change in baseline to week 4 is reported.
Measure: Mean (Standard Deviation); unit: pmol/min/μg of protein
Arm/Group | Active Stimulation (8) | Sham Stimulation (4), Active (4)
Number analyzed (Participants) | 4 | 4
pmol/min/μg of protein | 19.5 (27) | 6.47 (26.5)

4. Primary Outcome: Change in Mitochondrial Bioenergetics Measured by Basal Oxygen Consumption Rate at 8 Weeks (Basal Consumption)
Description: as for outcome 3
Time Frame: Assessed at baseline, week 4, and week 8. Change in baseline to week 8 is reported.
Measure: Mean (Standard Deviation); unit: pmol/min/μg of protein
Arm/Group | Active Stimulation (8) | Sham Stimulation (4), Active (4)
Number analyzed (Participants) | 4 | 1
pmol/min/μg of protein | 35.3 (7.6) | 31 (NA) — There were 4 subjects in the Sham group. All 4 had Week 0 Basal measures, but only 1 had Week 8 Basal measures. Therefore, there is only 1 subject with difference between Week 0 and Week 8 calculated, and thus there is no SD based on only 1 difference.

5. Primary Outcome: Change in Blood Cytokines Measured by TNF α Levels at 4 Weeks
Description: Blood will be analyzed to detect changes in protein cytokine TNF α levels, an indicator for inflammation.
Time Frame: Assessed at baseline, week 4, and week 8. Change in baseline to week 4 is reported.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Active Stimulation (8) | Sham Stimulation (4), Active (4)
Number analyzed (Participants) | 3 | 3
pg/mL | -0.237 (0.888) | -2.15 (3.80)

6. Primary Outcome: Change in Blood Cytokines Measured by TNF α Levels at 8 Weeks
Description: Blood will be analyzed to detect changes in protein cytokine TNF α levels, an indicator for inflammation
Time Frame: Assessed at baseline, week 4, and week 8. Change in baseline to week 8.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Active Stimulation (8) | Sham Stimulation (4), Active (4)
Number analyzed (Participants) | 3 | 1
pg/mL | -0.600 (3.17) | -1.35 (NA) — Only 1 participant in this group had Week 8 measures. Therefore, there is only 1 subject with difference between Week 0 and Week 8 calculated, and thus there is no SD based on only 1 difference.

7. Secondary Outcome: Change From Baseline in Functional Disability Inventory (Child and Adolescent)
Description: The Functional Disability Inventory (FDI) Child and Adolescent questionnaire will be used to assess change in symptoms. Participants will rank physical trouble or difficulty completing 15 different daily activities (Eating regular meals, Being at school all day, Walking up stairs, etc.) on a scale of 0-4 for each item (0-No trouble, 1- A Little Trouble, 2- Some Trouble, 3- A Lot of Trouble, 4- Impossible). Higher total scores indicate more difficulty functioning due to physical health, based on a sum score of each item. Sum score interpretation cutoffs include: No/Minimal Disability (0-12), Mild Disability (13-20), Moderate Disability (21-29) and Severe Disability (≥30).
Time Frame: Assessed at baseline, week 4, and week 8. Score changes from baseline to week 4 and baseline to week 8 are reported.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Active Stimulation (8) | Sham Stimulation (4), Active (4)
Number analyzed (Participants) | 4 | 4
Score on a scale
  Change from baseline to 4 weeks | -3.5 (10.2) | 0.75 (0.957)
  Change from baseline to 8 weeks | -2.50 (9.95) | 1.00 (1.00)

8. Secondary Outcome: Change From Baseline in Symptom Intensity Questionnaire
Description: Symptom Intensity Questionnaire score will be used to identify the most prominent 5 complaints, with intensity rated on a 10-point centimeter Likert scale. Participants write up to 5 of their most severe symptoms, and then rate those symptoms' severity from none (0) to worst you can possibly imagine (10) by placing a vertical line on the scale. Higher symptom ratings reflect higher symptom intensity & frequency. A 1-3 frequency level is a minimum level and indicates symptoms are occasional. A 4-6 frequency is a moderate level, meaning that symptoms are intermittent, coming and going. A 7-8 frequency is an indication that the symptoms are present more often than not but still not constant. A 9-10 frequency level is severe and indicates that symptoms are constant. The electronic data capture system's field validation used during the study automatically translated the participant-facing 0-10 slider scale placement into a score of 0-100, hence the reported mean values of over 10.
Time Frame: Assessed at baseline, week 4, and week 8. Changes per symptom score in baseline to week 4 and baseline to week 8 are reported.
Population: Only one participant reported a Symptom 5 Intensity at Week 4, as well as Symptoms 3, 4, and 5 Intensity at Week 8, therefore no Standard Deviation could be calculated for these results.
Measure: Mean (Standard Deviation); unit: Centimeters on a slider scale
Arm/Group | Active Stimulation (8) | Sham Stimulation (4), Active (4)
Number analyzed (Participants) | 4 | 4
Centimeters on a slider scale
  Symptom 1- Change from baseline to week 4 | 26 (29.7) | 6.75 (19.2)
  Symptom 2- Change from baseline to week 4 | 21 (27.4) | 4.25 (37.1)
  Symptom 3- Change from baseline to week 4 | -2.67 (12.1) | 26.7 (33.3)
  Symptom 4- Change from baseline to week 4 | -5 (14.1) | -9.5 (0.707)
  Symptom 5- Change from baseline to week 4: number analyzed (Participants) | 1 | 1
  Symptom 5- Change from baseline to week 4 | 20 (NA) — Only one participant reported symptom 5 intensity at both baseline & week 4. | -10 (NA) — Only one participant reported symptom 5 intensity at both baseline & week 4.
  Symptom 1- Change from baseline to week 8 | 78.7 (11) | 41.5 (33.1)
  Symptom 2- Change from baseline to week 8 | 60.5 (38.9) | 15.3 (18.6)
  Symptom 3- Change from baseline to week 8: number analyzed (Participants) | 1 | 1
  Symptom 3- Change from baseline to week 8 | 30 (NA) — Only one participant reported symptom 3 intensity at both baseline & week 8. | 15 (NA) — Only one participant reported symptom 3 intensity at both baseline & week 8.
  Symptom 4- Change from baseline to week 8: number analyzed (Participants) | 1 | 1
  Symptom 4- Change from baseline to week 8 | 65 (NA) — Only one participant reported symptom 4 intensity at both baseline & week 8. | 40 (NA) — Only one participant reported symptom 4 intensity at both baseline & week 8.
  Symptom 5- Change from baseline to week 8: number analyzed (Participants) | 1 | 1
  Symptom 5- Change from baseline to week 8 | 72 (NA) — Only one participant reported symptom 5 intensity at both baseline & week 8. | 70 (NA) — Only one participant reported symptom 5 intensity at both baseline & week 8.

9. Secondary Outcome: Change From Baseline in Pain Catastrophizing Scale (Child)
Description: The Pain Catastrophizing Scale Child form (PCS-C) will be completed by the participant. The PCS-C is a modification of the adult Pain Catastrophizing Scale for use in children, measuring pain-related cognitions and the dimensions of helplessness, rumination and magnification. Participants rate how strong their feelings are about pain on a 5 point scale (0- Not at all, 1- To a slight degree, 2- To a moderate degree, 3- To a great degree, 4- All the time). Sum scores range from 0-52. Higher scores indicate higher levels of pain catastrophizing. A total PCS score of 30 represents a clinically relevant level of catastrophizing.
Time Frame: Assessed at baseline, week 4, and week 8. Score change in baseline to week 8 is reported.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Active Stimulation (8) | Sham Stimulation (4), Active (4)
Number analyzed (Participants) | 4 | 4
Score on a scale | 2.5 (9.11) | -0.0667 (9.5)

10. Secondary Outcome: Change From Baseline in Revised Child Anxiety and Depression Scale
Description: The Revised Child Anxiety and Depression Scale (RCADS) assesses children grades 3 to 12 containing subscales assessing for symptoms of anxiety and depression. Participants rate frequency of occurrences described in the items on a 4 point scale (0- Never, 1- Sometimes, 2- Often, or 3- Always). Sum scores of anxiety/depression items were assessed.
  Depression items: score range 0-30 Anxiety items: score range 0-18
  Higher scores on both the depression & anxiety items indicate higher levels of depression & anxiety.
  Raw sum scores of both the depression & anxiety subscale items are translated to a T-score.
  T-scores below 65 represent low severity. T-scores between 65-70 represent medium severity and are on the borderline clinical threshold.
  T-scores above 70 represent high severity and are above the clinical threshold. A T-score of 50 indicates the population mean with a standard deviation of 10.
Time Frame: Assessed at baseline, week 4, and week 8. Changes in generalized anxiety & depression t-scores (translated from raw subscale scores) in baseline to week 4 and baseline to week 8 are reported.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Active Stimulation (8) | Sham Stimulation (4), Active (4)
Number analyzed (Participants) | 4 | 4
T-score
  Change from Baseline to 8 weeks- Major Depression Subscale | 0.75 (0.957) | -2.00 (3.00)
  Change from Baseline to 8 weeks- Generalized Anxiety Subscale | 1.00 (1.83) | 0.333 (0.577)

11. Secondary Outcome: Change From Baseline in Functional Disability Inventory (Parent)
Description: The Functional Disability Inventory (FDI) Parent questionnaire will be used to assess change in the participants symptoms as rated by the participants parent/guardian. Parents will rank their child's physical trouble or difficulty completing 15 different daily activities (Eating regular meals, Being at school all day, Walking up stairs, etc.) on a scale of 0-4 for each item (0-No trouble, 1- A Little Trouble, 2- Some Trouble, 3- A Lot of Trouble, 4- Impossible). Higher total scores indicate more difficulty functioning due to physical health, based on a sum score of each item. Sum score interpretation cutoffs include: No/Minimal Disability (0-12), Mild Disability (13-20), Moderate Disability (21-29) and Severe Disability (≥30).
Time Frame: Assessed at baseline, week 4, and week 8. Score changes from baseline to week 4 and baseline to week 8 are reported.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Active Stimulation (8) | Sham Stimulation (4), Active (4)
Number analyzed (Participants) | 4 | 4
Score on a scale
  Change from baseline to week 4 | -6.25 (5.12) | -2.5 (1.73)
  Change from baseline to week 8 | -3.67 (9.29) | -8 (7.96)

12. Secondary Outcome: Change From Baseline in Pain Catastrophizing Scale (Parent)
Description: The Pain Catastrophizing Scale Parent form (PCS-P) will be completed by the parent or guardian of the participant. The PCS-P is a proxy questionnaire to the PCS-C, measuring the feelings the parent has when their child is in pain. Parents rate how strongly they feel when their child is in pain on a 5 point scale (0- Not at all, 1- To a slight degree, 2- To a moderate degree, 3- To a great degree, 4- All the time). Sum scores range from 0-52. Higher scores indicate higher levels of pain catastrophizing. A total PCS score of 30 represents a clinically relevant level of catastrophizing.
Time Frame: Assessed at baseline, week 4, and week 8. Score change from baseline to week 8 is reported.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Active Stimulation (8) | Sham Stimulation (4), Active (4)
Number analyzed (Participants) | 4 | 4
Score on a scale | -5.67 (7.51) | -3.0 (9.42)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 2 months.
Description: Participants contacted the study team to report adverse events.
Groups:
- Active Stimulation for 4 Weeks (Following Sham Stimulation); Sham Stimulation for 4 Weeks: Participants will receive sham therapy via inactive TENS unit for 4 weeks, followed by active auricular microstimulation via TENS for 4 weeks.
  Under guidance from the study team, participants will self-administer the TENS therapy for two 1-hour periods a day for 8 weeks (4 weeks of therapy with inactive TENS, 4 weeks with active TENS).
  Transcutaneous Electrical Nerve Stimulation (TENS): Active Transcutaneous Auricular Microstimulation delivered by TENS device
  Sham Transcutaneous Electrical Nerve Stimulation: Sham therapy will be delivered by applying the TENS device with non-conductive electrodes so that no microstimulation is delivered.
  Participants in this group received both sham and active stimulation.
Arm/Group | Active Stimulation (8) | Active Stimulation for 4 Weeks (Following Sham Stimulation) | Sham Stimulation for 4 Weeks
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 1/5 | 0/5 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Stimulation (8) (N=5) | Active Stimulation for 4 Weeks (Following Sham Stimulation) (N=5) | Sham Stimulation for 4 Weeks (N=5)
Gastrointestinal Symptoms (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Subject used TENS device for the first time 4/8/21 and woke up 4/9/21 with nausea, stomach pain, diarrhea and hiccups. Symptoms did not improve after 5 days, so subject was withdrawn at PI discretion and referred for GI follow-up. Unrelated to TENS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-17): https://cdn.clinicaltrials.gov/large-docs/00/NCT04247100/Prot_SAP_000.pdf